CLINICAL TRIAL: NCT01993017
Title: Depression Screening RCT in ACS Patients: Quality of Life and Cost Outcomes
Brief Title: Comparison of Depression Identification After Acute Coronary Syndrome: Quality of Life and Cost Outcomes
Acronym: CODIACSQoL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Duke University (Other); HealthPartners Institute (Other); Kaiser Foundation Research Institute (Other)
Responsible Party: Principal Investigator, Ian Kronish, Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: AAAK9253; 1R01HL114924 (NIH)
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Acute Coronary Syndrome; Depressive Symptoms
Keywords: Acute Coronary Syndrome; Depressive Symptoms
MeSH Terms: conditions — Acute Coronary Syndrome; Depression | interventions — Cognitive Behavioral Therapy; Antidepressive Agents; Sertraline; Bupropion; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AHA Depression Screen & Treat (Experimental): Participants randomized to this arm will complete the Depressive symptom screener (8-item Patient Health Questionnaire, PHQ-8) after randomization. Those with clinically significant score (>=10) will be offered treatment. Treatment will be delivered according to participant preference, and will be managed according to "stepped care". Stepped care includes, a) participant preference for either brief, cognitive behavioral therapy (CBT), delivered centrally by telephone, or antidepressant medication managed at the local site, or both, or neither, and b) review of progress at approximately 2-month intervals, with "stepping up" of care if sufficient progress is not being realized.
  Interventions: Other: Cognitive Behavioral Therapy (CBT); Drug: Antidepressant Medication; Other: Depressive symptom screener
- Depression Screen & Notify Arm Type : (Active Comparator): Participants randomized to this arm will complete the depressive symptom screener (8-item Patient Health Questionnaire, PHQ-8) after randomization. Those with clinically significant score (>=10) will have a letter sent to their primary care provider about their positive screen for depressive symptoms, with subsequent actions at the provider's discretion.
  Interventions: Other: Standard Care; Other: Depressive symptom screener
- No Depression Screen (Placebo Comparator): Participants randomized to this arm will not complete a PHQ-8 assessment at randomization, and so will not be screened for depressive symptoms.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Cognitive Behavioral Therapy (CBT) — The main intervention is the impact of screening on quality of life and health care costs. CBT is provided only if depressive symptoms are detected and participant prefers this type of treatment.
  CBT will be centrally telephone-administered by a trained CBT treatment specialist. The treatment specialist will work with local team members throughout a participant's involvement in the study, and will closely follow each participant until he or she has reached a requisite level of improvement .
  Other Names: Problem Solving Therapy (PST)
  Arms: AHA Depression Screen & Treat
Drug: Antidepressant Medication — The main intervention is the impact of screening on quality of life and health care costs. Antidepressant Medication is provided only if depressive symptoms are detected and patient prefers this type of treatment.
  Antidepressants should be started at the lowest dose, but should be adjusted upward to be within the therapeutic range within 1 week, with further adjustment higher in the therapeutic range possible at 3-4 weeks. Dosage of the first medication selected will be in the therapeutic range by 3 weeks of the initial step, as tolerated.
  Other Names: Sertraline; Bupropion
  Arms: AHA Depression Screen & Treat
Other: Standard Care — Participants will receive standard care from either their primary care provider (PCP), or PCP-referred mental health provider in one of the arms, IF depressive symptoms are detected.
  Arms: Depression Screen & Notify Arm Type :
Other: Depressive symptom screener — 8-item Patient Health Questionnaire, PHQ-8
  Other Names: PHQ-8
  Arms: AHA Depression Screen & Treat; Depression Screen & Notify Arm Type :
Other: No intervention
  Arms: No Depression Screen

SUMMARY:
The purpose of this study is to examine, in a randomized controlled trial, the benefits and costs of the American Heart Association's (AHA) advisory for depression screen and treatment of post-acute coronary syndrome patients.

DETAILED DESCRIPTION:
Patients with an acute coronary syndrome (ACS) and comorbid depression have a 2-fold higher risk for recurrent ACS and mortality, worse quality of life, and higher costs of care than nondepressed ACS patients. The strength of these observational findings prompted the American Heart Association (AHA) to advise that routine depression screening for ACS patients and referral for depression diagnosis and treatment as indicated occur. Unfortunately, there are no randomized controlled trials (RCT) to inform this potentially expensive screening recommendation. Additionally, screening guidelines/advisories in the absence of RCT evidence have recently been extensively criticized (and withdrawn). This poses a serious dilemma for clinicians, health care systems, and for health care policy leaders. A RCT is urgently needed to provide evidence for these different constituents about the costs and benefits of the AHA depression screen and treat algorithm.

Two critical gaps in knowledge must be filled to determine if public health would be improved by the AHA strategy for depression screening in post-ACS patients: 1) Does this strategy improve quality-adjusted life years for patients with a recent ACS 2) Is the cost of providing depression screening and any type of depression treatment within the acceptable and typical amounts reimbursed for health care services? Our specific aim is to determine the quality-adjusted life year benefits and health care costs of following the AHA's advisory for depression screening and then referral for further diagnosis and treatment in post-ACS patients, if depression is found. To accomplish this aim, we will randomize patients from four different, geographically diverse health care systems to three different groups: 1) to the AHA depression screen and treat if depression is found algorithm (screen and treat intervention group) or: 2) to be screened and a primary care provider notified (screen and notify intervention group) or: 3) to receive no depression screening (control group). Health-related quality of life, depressive symptoms, and costs will be obtained from all patients, so that the benefits and the costs of these three different depression screening strategies can be compared.

ELIGIBILITY:
Inclusion Criteria:

* With a documented acute coronary syndrome (ACS) within the past 2-12 months
* Over the age of 21 years
* Has access to a phone

Exclusion Criteria:

Medical Exclusions:

* Terminal illness (life expectancy <1 year as determined by physician/medical record) defined as, but not limited to:
* NYHA class IV, ACC class D CHF requiring inotropes or mechanical assist devices or critical aortic stenosis without plan for correction
* End-stage COPD/emphysema
* Advanced cirrhosis with encephalopathy, varices, severe ascites
* Severe rheumatologic diseases requiring frequent hospitalizations, and multiple cytotoxic agents and/or disease modifying drugs
* Metastatic pancreatic, esophageal, colorectal or stomach cancer
* Metastatic sarcoma, ovarian, melanoma or renal cell cancer
* Metastatic breast cancer with multiple recurrences despite treatment
* Advanced CNS malignancies
* Recurrent hematologic malignancies with multiple recurrences despite treatment
* Persistent AIDS, untreated or treated

Psychiatric Exclusions:

* History of major depression
* Currently receiving depression treatment
* Dementia
* History of bipolar disorder
* History of psychosis
* History of suicide attempt or self-inflicted injuries
* Current alcohol or substance abuse

Other Exclusions:

* Non-English and non-Spanish speaking

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1501 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Kronish, MD, MPH, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - Health Partners institute for Research and Education, Bloomington, Minnesota
  - Columbia University Irving Medical Center, New York, New York
  - Duke University, Henderson, North Carolina
  - Kaiser Foundation Research Institute, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
A deidentified data set and study materials will be provided upon request by other researchers.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Starting in January 2021
Access Criteria: Contact the study PI with data requests

REFERENCES:
- [Background] Moise N, Davidson KW, Cheung YKK, Clarke GN, Dolor RJ, Duer-Hefele J, Ladapo JA, Margolis KL, St Onge T, Parsons F, Retuerto J, Schmit KM, Thanataveerat A, Kronish IM. Rationale, design, and baseline data for a multicenter randomized clinical trial comparing depression screening strategies after acute coronary syndrome: The comparison of depression identification after acute Coronary Syndromes-Quality of Life and Cost Outcomes (CODIACS-QOL) trial. Contemp Clin Trials. 2019 Sep;84:105826. doi: 10.1016/j.cct.2019.105826. Epub 2019 Aug 13. PMID 31419605
- [Result] Kronish IM, Moise N, Cheung YK, Clarke GN, Dolor RJ, Duer-Hefele J, Margolis KL, St Onge T, Parsons F, Retuerto J, Thanataveerat A, Davidson KW. Effect of Depression Screening After Acute Coronary Syndromes on Quality of Life: The CODIACS-QoL Randomized Clinical Trial. JAMA Intern Med. 2020 Jan 1;180(1):45-53. doi: 10.1001/jamainternmed.2019.4518. PMID 31633746
- [Result] Ladapo JA, Davidson KW, Moise N, Chen A, Clarke GN, Dolor RJ, Margolis KL, Thanataveerat A, Kronish IM. Economic outcomes of depression screening after acute coronary syndromes: The CODIACS-QoL randomized clinical trial. Gen Hosp Psychiatry. 2021 Jul-Aug;71:47-54. doi: 10.1016/j.genhosppsych.2021.04.001. Epub 2021 Apr 3. PMID 33933921

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: November 1, 2013 to March 31, 2017
  Recruitment sites: HealthPartners (Minneapolis, Minnesota), Duke University Health System (Durham, North Carolina), Kaiser Permanente Northwest (Portland, Oregon), and New York-Presbyterian/Columbia University Irving Medical Center (New York, New York)
Pre-assignment Details: 1 participant withdrew consent soon after randomization, and this participant's data was excluded from the study.
Groups:
- AHA Depression Screen, Notify & Treat: Participants randomized to this arm will complete the Depressive symptom screener (8-item Patient Health Questionnaire, PHQ-8) after randomization. Those with clinically significant score (>=10) will be offered treatment. Treatment will be delivered according to participant preference, and will be managed according to "stepped care". Stepped care includes, a) participant preference for either brief, type of cognitive behavioral therapy (CBT) called problem-solving therapy (PST), delivered centrally by telephone, or antidepressant medication managed at the local site, or both, or neither, and b) review of progress at approximately 2-month intervals, with "stepping up" of care if sufficient progress is not being realized.
- Depression Screen & Notify: Participants randomized to this arm will complete the depressive symptom screener (8-item Patient Health Questionnaire, PHQ-8) after randomization. Those with clinically significant score (>=10) will have a letter sent to their primary care provider about their positive screen for depressive symptoms, with subsequent actions at the provider's discretion.
  Standard Care: Participants will receive standard care from either their primary care provider (PCP), or PCP-referred mental health provider in one of the arms, IF depressive symptoms are detected.
  Depressive symptom screener: 8-item Patient Health Questionnaire, PHQ-8
- No Depression Screen: Participants randomized to this arm will not complete a PHQ-8 assessment at randomization, and so will not be screened for depressive symptoms.
  No intervention
Period: Overall Study
Arm/Group | AHA Depression Screen, Notify & Treat | Depression Screen & Notify | No Depression Screen
Started | 499 | 501 | 500
Completed | 393 | 411 | 421
Not Completed | 106 | 90 | 79
Not completed — Death | 23 | 26 | 18
Not completed — Could not be contacted | 43 | 42 | 38
Not completed — Dropped out | 19 | 6 | 11
Not completed — Other reasons | 17 | 11 | 7
Not completed — Ineligible after randomization | 4 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- AHA Depression Screen, Notify & Treat: Participants randomized to this arm will complete the Depressive symptom screener (8-item Patient Health Questionnaire, PHQ-8) after randomization. Those with clinically significant score (>=10) will be offered treatment. Treatment will be delivered according to participant preference, and will be managed according to "stepped care". Stepped care includes, a) participant preference for either a type of brief, cognitive behavioral therapy (CBT) called problem solving therapy (PST), delivered centrally by telephone, or antidepressant medication managed at the local site, or both, or neither, and b) review of progress at approximately 2-month intervals, with "stepping up" of care if sufficient progress is not being realized.
- Total: Total of all reporting groups
Arm/Group | AHA Depression Screen, Notify & Treat | Depression Screen & Notify | No Depression Screen | Total
Number analyzed (Participants) | 499 | 501 | 500 | 1500
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (11.3) | 65.8 (11.7) | 65.8 (11.7) | 65.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 137 | 145 | 424
  Male | 357 | 364 | 355 | 1076
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 82 | 88 | 74 | 244
  Not Hispanic or Latino | 406 | 402 | 410 | 1218
  Unknown or Not Reported | 11 | 11 | 16 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 353 | 368 | 359 | 1080
  Black | 47 | 37 | 46 | 130
  Other | 92 | 82 | 85 | 259
  Refused or unknown | 7 | 14 | 10 | 31
Region of Enrollment [Number; unit: participants]
  United States | 499 | 501 | 500 | 1500
PHQ-8 Score >= 10 [Count of Participants; unit: Participants] — Population: PHQ-8 data were not collected at Baseline in the "No Depression Screen" Arm/Group).
  Participants
    number analyzed (Participants) | 494 | 501 | 0 | 995
    (all) | 38 | 33 |  | 71

OUTCOME MEASURES:

1. Primary Outcome: Quality-Adjusted Life Years (QALYs)
Description: Change in QALYs from baseline through 18 months. QALYs are a generic measure of disease burden, including both the quality and the quantity of life lived. One QALY equates to one year in perfect health. To measure change in QALYs, utility scores [an overall assessment of well-being on a scale from 0 (death) to 1 (perfect health)], were estimated using the Short Form-6 dimension, with scores derived from responses to the 12-Item Short-Form Health Survey, version 2, at baseline and 6, 12, and 18 months. QALYs for the period from baseline to 18 months were then calculated as the area under the curve by linearly interpolating the utility scores at the 4 assessments. Change in QALYs was then obtained by subtracting the baseline QALY from the observed QALY for an 18-month period, where baseline QALY was calculated under the assumption that the baseline utility score remained constant during the 18-month period.
Time Frame: Baseline, 6, 12 and 18 months
Measure: Mean (Standard Deviation); unit: quality-adjusted life years (QALYs)
Arm/Group | AHA Depression Screen, Notify & Treat | Depression Screen & Notify | No Depression Screen
Number analyzed (Participants) | 499 | 501 | 500
quality-adjusted life years (QALYs) | -0.06 (0.20) | -0.06 (0.20) | -0.06 (0.18)
Statistical Analysis 1: Comparison: AHA Depression Screen, Notify & Treat vs Depression Screen & Notify vs No Depression Screen; We determined that a sample size per group of 500, assuming 5% loss to follow-up, would yield 80% power for a 2-sided t test at the 5% level. These calculations were based on an assumed SD for QALYs of 0.17, expected prevalence of screening-detected depression of 20%, and assumed net improvement in QALYs of 0.155 over 18 months for individuals with depression who received treatment for depression in the Screen, Notify, and Treat group; Test type: Superiority; p = 0.98, ANOVA — A 2-step gatekeeping test procedure was used. An omnibus F test using ANOVA comparing the 3 groups was first performed. Pairwise comparisons using a 2-sided t test at 5% nominal significance were planned only if the omnibus F test had a P value <.05

2. Secondary Outcome: Depression-free Days
Description: Depression-free days from baseline through 18 months post-randomization
Time Frame: Baseline through 18 months
Measure: Mean (Standard Deviation); unit: cumulative depression-free days
Arm/Group | AHA Depression Screen, Notify & Treat | Depression Screen & Notify | No Depression Screen
Number analyzed (Participants) | 499 | 501 | 500
cumulative depression-free days | 343.1 (179.0) | 351.3 (175.0) | 339.0 (176.6)

3. Secondary Outcome: Cost of Health Care Utilization
Description: Total cost of health care utilization from baseline through 18 months post-randomization
Time Frame: Baseline through 18 months
Measure: Mean (Standard Error); unit: US dollars
Arm/Group | AHA Depression Screen, Notify & Treat | Depression Screen & Notify | No Depression Screen
Number analyzed (Participants) | 499 | 501 | 500
US dollars | 6745 (358) | 6204 (332) | 7440 (501)

ADVERSE EVENTS:
Time Frame: 18 months
Description: Serious Adverse Events and mortality were assessed in all participants.
  Other Adverse Events were assessed using a self-report instrument at 6-mo, 12-mo, and 18-mo. As not all participants were reached to complete this questionnaire, fewer participants were assessed for Other Adverse Events than for Serious Adverse Events and mortality. Also, the number of participants who were assessed for Other Adverse Events varies according to the time period of assessment.
Arm/Group | AHA Depression Screen, Notify & Treat | Depression Screen & Notify | No Depression Screen
All-Cause Mortality (participants affected / at risk) | 23/499 | 26/501 | 18/500
Serious Adverse Events (participants affected / at risk) | 0/499 | 0/501 | 0/500
Other Adverse Events (participants affected / at risk) | 386/450 | 398/455 | 399/458
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | AHA Depression Screen, Notify & Treat (N=450) | Depression Screen & Notify (N=455) | No Depression Screen (N=458)
Any bleeding at 6 mo (Blood and lymphatic system disorders) | 61 | 51 | 72/457 — Self-report of any bleeding
Increased appetite at 6 mo (Psychiatric disorders) | 83 | 84 | 91/457 — Self-report of increased appetite
Decreased appetite at 6 mo (Psychiatric disorders) | 72 | 74 | 76/457 — Self-report of decreased appetite
Drowsiness at 6 mo (Psychiatric disorders) | 218 | 212 | 217 — Self-report of drowsiness
Gastrointestinal upset at 6 mo (Gastrointestinal disorders) | 128 | 116/454 | 112/457 — Self-report of gastrointestinal upset
Any bleeding at 12 mo (Blood and lymphatic system disorders) | 51/423 | 50/429 | 50/427
Increased appetite at 12 mo (Psychiatric disorders) | 71/423 | 77/431 | 76/427
Decreased appetite at 12 mo (Psychiatric disorders) | 63/423 | 65/431 | 76/427
Drowsiness at 12 mo (Psychiatric disorders) | 179/423 | 187/431 | 198/427
Gastrointestinal upset at 12 mo (Gastrointestinal disorders) | 95/423 | 95/431 | 107/427
Any bleeding at 18 mo (Blood and lymphatic system disorders) | 40/394 | 45/410 | 40/419
Increased appetite at 18 mo (Psychiatric disorders) | 76/394 | 62/410 | 60/418
Decreased appetite at 18 mo (Psychiatric disorders) | 53/394 | 45/410 | 62/419
Drowsiness at 18 mo (Psychiatric disorders) | 152/394 | 177/410 | 171/419
Gastrointestinal upset at 18 mo (Gastrointestinal disorders) | 98/394 | 99/410 | 100/418

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT01993017/Prot_002.pdf
  • Statistical Analysis Plan (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT01993017/SAP_001.pdf